CLINICAL TRIAL: NCT00917501
Title: Neurochemical Effects of Omega-3 Fatty Acids in Adolescents at Risk for Mania
Acronym: R34
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Cincinnati (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Robert McNamara, Professor, University of Cincinnati
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Del/McNa OMega 3; MH083924
Record Dates: First submitted 2009-06-08; First posted 2009-06-10 (Estimated); Results first posted 2016-06-09 (Estimated); Last update posted 2019-11-13 (Actual); Status verified 2019-10

CONDITIONS: Mania
Keywords: Mania; Adolescents at risk for Mania
MeSH Terms: conditions — Mania | interventions — Docosahexaenoic Acids; Fish Oils; Olive Oil

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): Placebo to the Omega-3 given in other group taken twice a day.
  Interventions: Drug: Placebo
- Omega 3 (Active Comparator): Individual omega-3 capsules contain 400 mg EPA and 200 mg DHA & will be taken twice a day.
  Interventions: Drug: OMega 3

INTERVENTIONS:
Drug: OMega 3 — Individual omega-3 capsules contain 400 mg EPA and 200 mg DHA taken twice a day
  Other Names: Fish oil
  Arms: Omega 3
Drug: Placebo — Placebo given twice a day which will be compared to Omega 3
  Other Names: Olive oil
  Arms: Placebo

SUMMARY:
The purpose of this study is to see if taking a substance called omega-3 fatty acids is effective, safe, and well-tolerated for treating adolescents with major depressive disorder (also called simply "depression" or "clinical depression"). Another purpose of this study is to see how much omega-3 fatty acids are in a patient's blood and if that makes the patient more or less likely to develop mania (i.e. periods of irritability or extreme silliness accompanied by decreased need for sleep, risky behaviors, feeling like the patient has special abilities, inability to sit still, and rapid speech) in the future. Yet another purpose of this study is to see how taking omega-3 fatty acids affect brain scans. Omega-3 fatty acids are not United States Food and Drug Administration (FDA)-approved to treat depression in adults or in children and adolescents.

Omega-3 fatty acids can only be obtained through diet, most often from fish and other sea foods, though they are also found in other food sources such as flax seed. Omega-3 fatty acids have been shown to play a role in affecting brain chemicals responsible for regulating mood and have been found to reduce symptoms of depression in medicated-patients with major depressive disorder.

By completing this study, the investigators hope to better understand who benefits from treatment, why they do or do not respond to medications, and who is at greater risk for developing further mental illness. With this information, the investigators hope to be able to improve treatment and outcome in people with major depressive disorder.

DETAILED DESCRIPTION:
A. Specific Aims: (1) To collect pilot data regarding the efficacy, safety, and tolerability of omega-3 fatty acid supplementation for the treatment of adolescents with active depressive symptoms and a high risk for developing mania (i.e. the patient has a bipolar parent and meet DSM-IV-TR criteria for major depressive disorder). (2) To use proton magnetic resonance spectroscopy (1H MRS) (i.e. prefrontal neurochemistry) and red blood cell (RBC) omega-3 fatty acid levels to examine potential mediators of treatment response to omega-3 fatty acids in adolescents with a high risk for mania.

ELIGIBILITY:
Inclusion Criterion:

* Ages 10-21 years old.
* At least one biological parent with bipolar I disorder.
* Meets DSM-IV-TR 80 criteria for major depressive disorder (MDD or Depressive Disorder NOS at screening as determined by the Washington University at St. Louis Kiddie Schedule for Affective Disorders and Schizophrenia, WASH-U-KSADS;81
* Childhood Depression Rating Scale-Revised Version40,41(CDRS-R) scores greater than or equal to 40 at screening and baseline.
* Fluent in English.
* Provision of written informed consent/assent as previously described.
* Agrees to use one of the following method of birth control: complete abstinence from sexual intercourse, barrier (diaphragm or condom), or oral/injectable contraceptive.

Exclusion Criterion:

* Contraindication to an MRI scan (e.g., metal clips, braces or claustrophobia).
* Mood symptoms resulting from acute medical illness or acute intoxication or withdrawal from drugs or alcohol as determined by careful medical evaluation or rapid symptom resolution.
* Psychotic symptoms (i.e., hallucinations or delusions).
* Any lifetime history of a manic or hypomanic episode.
* Any lifetime diagnosis of bipolar disorder not otherwise specified (NOS) or cyclothymia or a current diagnosis of depressive disorder NOS. A current diagnosis of dysthymia will not be exclusionary, if the adolescent also has a current diagnosis of MDD.
* A history of a major medical (e.g. diabetes) or neurological illness, laboratory abnormalities, or a significant episode (> 10 minutes) of loss of consciousness that could influence the MRS results, as determined by a study physician.
* Any history of alcohol or drug dependence (nicotine dependence is permitted).
* Allergy to shellfish or seafood.
* Mental retardation (IQ<70) as determined by the Wechsler Abbreviated Scale of Intelligence (WASI), administered by a research coordinator who is a trained psychometrician.
* A positive serum pregnancy test or lactating.
* A history of intolerance, hypersensitivity or non-response to omega-3 fatty acids.
* Any history of a hematological disorder in themselves or a first-degree relative, since omega-3 fatty acids may be associated with anti-coagulant effects.
* Concomitant use of medications with anticoagulant effects (e.g. aspirin).
* A lithium or valproate serum level of >0.4 mEq/L and 30 mg/L, respectively at baseline.
* Use of antipsychotics, other mood stabilizers, stimulants (if opting to discontinue), or atomoxetine within 72 hours (aripiprazole within two weeks will be exclusionary because of its long half-life) or antidepressants within 5 days (fluoxetine within one month will be exclusionary because of its long half-life). Patients treated with a depot antipsychotic within one dosing interval of baseline will be excluded. Subjects diagnosed with ADHD and taking a stable dose of stimulants for the previous month will be permitted to continue if it is determined necessary by subject, primary caregiver, and treating clinician report in conjunction with the study physician.
* Concomitant use of other psychotropic medications or medications with central nervous system (CNS) effects within 5 half-lives from baseline MRI scan or prior treatment with a medication with CNS effects that requires more than 5 days of a screening period.
* Any psychiatric symptom that requires admission to an inpatient psychiatric hospital, as determined by a study physician.
* Any initiated psychotherapy within 2 months prior to the screening visit, or plans to initiate psychotherapy during study participation. Adolescents who present with their current depressive episode despite longer-term psychotherapy (i.e., >2 months) may be included. For participants who enter the study on psychotherapy, the type and frequency of therapy will remain constant during the study.

Ages: 10 Years to 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 55 (Actual)
Dates: Start 2009-06; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Melissa DelBello, MD, Principal Investigator — University of Cincinnati; Robert McNamara, PhD, Principal Investigator — University of Cincinnati
Locations (1):
- University of Cincinnati, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Olive oil - 3 capsules/day
- Omega-3: Fish oil - 3 capsules/day
Period: Overall Study
Arm/Group | Placebo | Omega-3
Started | 29 | 26
Completed | 21 | 21
Not Completed | 8 | 5
Not completed — Lost to Follow-up | 4 | 1
Not completed — Withdrawal by Subject | 3 | 1
Not completed — Lack of Efficacy | 1 | 2
Not completed — trouble swollowing capsules | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Omega-3 | Total
Number analyzed (Participants) | 29 | 26 | 55
Age, Continuous [Mean (Standard Deviation); unit: Years] | 13.4 (3.3) | 13 (4.5) | 13.2 (3.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 21 | 45
  Male | 5 | 5 | 10
Region of Enrollment [Number; unit: participants]
  United States | 29 | 26 | 55

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Depression Symptom Severity at 12 Weeks
Description: Change in Children's Depression Rating Scale-revised (CDRS-R) Total Score from Baseline to 12 weeks CDRS-R score ranges from 17 (i.e., not depressed) to 113 (i.e., severe depression)
Time Frame: Baseline and 12 weeks
Measure: Mean (Standard Deviation); unit: Total score on CDRS-R
Arm/Group | Placebo | Omega-3
Number analyzed (Participants) | 29 | 26
Total score on CDRS-R | 18 (9.7) | 17.7 (11)

ADVERSE EVENTS:
Arm/Group | Placebo | Omega-3
Serious Adverse Events (participants affected / at risk) | 0/29 | 0/26
Other Adverse Events (participants affected / at risk) | 0/29 | 8/26
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=29) | Omega-3 (N=26)
Muscle Cramps (General disorders) | 0 (0) | 8 (10)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No